CLINICAL TRIAL: NCT03987568
Title: To Characterize Tumor Hypoxia by Magnetic Resonance Imaging in African American and Caucasian Prostate Cancer Patients
Brief Title: Characterize Tumor Hypoxia by Magnetic Resonance Imaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues in reserving MRI scanner
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00059037; WFBCCC 03319 (Other: Wake Forest Baptist Comprenhensive Cancer Center); P30CA012197 (NIH); NCI-2019-04690 (Other: National Cancer Institute)
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer; Prostate Tumor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (MRI biospecimen collection) (Experimental): Patients undergo MRI over 15 minutes before standard of care surgery. Patients also undergo collection of blood samples during MRI and at the time of surgery.
  Interventions: Other: Blood draws; Diagnostic Test: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Other: Blood draws — Blood draws at two specified timepoints - the first is during the MRI and the second is scheduled during participant's prostatectomy.
Diagnostic Test: Magnetic resonance imaging (MRI) — At the beginning of study magnetic resonance imaging MRI will be completed.

SUMMARY:
The purpose of this research study is to measure the hypoxia (low oxygen condition) in prostate cancers and its effect in survival. In this study, investigators will assess hypoxia by magnetic resonance imaging (MRI) and create a hypoxia score. Investigators will study the hypoxia score and how it correlates (if any) to the disease aggressiveness as well as its effect on the treatment outcomes.

DETAILED DESCRIPTION:
Primary Objective(s):

* To assess hypoxia in primary prostate tumors by magnetic resonance imaging.
* To correlate hypoxic score with disease aggressiveness (proliferation biomarkers' expression).

Secondary Objective(s):

* To correlate hypoxic score with ExoHypoxic concentration in plasma of same patient.
* To correlate hypoxic score with fatty acid synthase (FASN) expression.

ELIGIBILITY:
Inclusion Criteria:

* The minimum age for this study is men 40 years and older. Prostate cancer mainly affects men over the age of 40.
* Patients with Caucasian and African American race
* Patients with pathology-proven prostate cancer (Gleason 6 or higher)
* Patients who have not yet undergone therapy (systemic drugs, radiation, or prostatectomy)
* Patients who will have a radical prostatectomy as standard of care.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Patients who have already received some form of treatment or are not planning to undergo radical prostatectomy for treatment.
* Patients with any other cancer along with prostate cancer.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Differences in Tumor Hypoxia Scores Between Subgroups | 30 days
  Using MRI parameters including apparent diffusion coefficient and fractional blood value four race/score combination groups (African-Americans with Gleason score 6; African-Americans with Gleason score greater than or equal to 7; Caucasians with Gleason score 6; and Caucasian with Gleason score greater than or equal to 7) to calculate the correlation coefficients estimates between hypoxic scores using Pearson correlation coefficient and Spearman's rank correlation coefficient.
Number of Biomarkers Expressed | 30 days
  Expression of proliferation biomarkers (Ki-67 and PCNA) to calculate the correlation coefficients estimates between expression of proliferation biomarkers using Pearson correlation coefficient and Spearman's rank correlation coefficient.

SECONDARY OUTCOMES:
ExoHypoxic Concentrations in Plasma | 30 days
  The associations between hypoxic score and candidate biomarkers for ExoHypoxic concentration (number per milliliter plasma) will be estimated using partial Spearman's rank correlation coefficient where the race/score combination groups are adjusted.
Number of Fatty Acid Synthase Expressions in Prostate Cancer and ExoHypoxic Concentrations | 30 days
  The associations between hypoxic score and fatty acid synthase expression will be estimated using partial Spearman's rank correlation coefficient where the race/score combination groups are adjusted.

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Deep, Ph.D, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No